CLINICAL TRIAL: NCT07225842
Title: The Bridging Antiplatelet Therapy With Cangrelor 2 (BRIDGE 2) Study: A Pilot Prospective Cohort, Pharmacodynamic Study of Tailored Cangrelor Bridging Dosing Regimens
Brief Title: The Bridging Antiplatelet Therapy With Cangrelor 2 Study
Acronym: BIRDGE 2
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB202500991
Record Dates: First submitted 2025-11-06; First posted 2025-11-10 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-09

CONDITIONS: Coronary Arterial Disease (CAD)
Keywords: coronary artery disease; cangrelor; bridge
MeSH Terms: conditions — Coronary Artery Disease | interventions — cangrelor

STUDY DESIGN:
Intervention Model Description: After providing informed consent, eligible patients will undergo a baseline evaluation of PRU levels by means of the VerifyNow system. The research study team will perform the PRU assessment in the cardiovascular research lab as this is considered a research only assessment and is not currently performed as standard of care. Patients with PRU levels ≤208 will undergo cangrelor dose reduction to 0.50 mcg/kg/min, while patients with PRU levels >208 will undergo dose increase to 1.0 mcg/kg/min. At 2 to 12 hours after dose titration, blood samples will be collected for further PD assessment of platelet reactivity. Patients with PRU values >208 will undergo dose increase by 0.25 mc/kg/min up to a maximum of 1.5 mcg/kg/min until a PRU below 208 is achieved, while patients with PRU levels <85 will undergo dose reduction to 0.25 mcg/kg/min, being the lowest possible administration rate allowed during the study period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Platelet function-guided cangrelor titration (Experimental): Patients with PRU levels ≤208 will undergo cangrelor dose reduction to 0.50 mcg/kg/min, while patients with PRU levels >208 will undergo dose increase to 1.0 mcg/kg/min. At 2 to 12 hours after dose titration, blood samples will be collected for further PD assessment of platelet reactivity. Patients with PRU values >208 will undergo dose increase by 0.25 mc/kg/min up to a maximum of 1.5 mcg/kg/min until a PRU below 208 is achieved, while patients with PRU levels <85 will undergo dose reduction to 0.25 mcg/kg/min, being the lowest possible administration rate allowed during the study period. Titration will be performed at 3 time points: baseline (while on 0.75 mcg/kg/min before dose titration); between 2 and 12 hours following dose titration; daily (at the same time for the second dose) for up to a maximum of 3 samples after dose titration.
  Interventions: Drug: Cangrelor

INTERVENTIONS:
Drug: Cangrelor — Patients with PRU levels ≤208 will undergo cangrelor dose reduction to 0.50 mcg/kg/min, while patients with PRU levels >208 will undergo dose increase to 1.0 mcg/kg/min. At 2 to 12 hours after dose titration, blood samples will be collected for further PD assessment of platelet reactivity. Patients with PRU values >208 will undergo dose increase by 0.25 mc/kg/min up to a maximum of 1.5 mcg/kg/min until a PRU below 208 is achieved, while patients with PRU levels <85 will undergo dose reduction to 0.25 mcg/kg/min, being the lowest possible administration rate allowed during the study period. Titration will be performed at 3 time points: baseline (while on 0.75 mcg/kg/min before dose titration); between 2 and 12 hours following dose titration; daily (at the same time for the second dose) for up to a maximum of 3 samples after dose titration.

SUMMARY:
The primary aim of this study is to determine rates of patients with optimal platelet reactivity range, defined as PRU levels between 85 and 208, when using a (PFT)-guided titration of cangrelor infusion rate (cangrelor titration) compared to 0.75 mcg/kg/min (standard-dose infusion) for bridging.

DETAILED DESCRIPTION:
The proposed investigation is a prospective, single-arm, open-label PD study in patients that are admitted to UF Health Jacksonville with established coronary artery disease. These patients will be awaiting a coronary intervention in the cardiac cath lab or a coronary artery bypass graft in the operating room and have received at least a two-hour infusion of cangrelor as standard of care for bridging at 0.75 mcg/kg/min (standard-dose infusion).The typical wait time for the patient's aforementioned procedure/surgery is 5 days or more and the study schedule will not interfere with the typical clinical processes. If the patient's procedure or surgery is re-scheduled to an earlier than expected time, then the study procedures will stop and will not delay the patient's standard of care procedure/surgery. . Patients will be recruited from the inpatient units of the institution and screened by the Cardiology Research staff, who will verify that all candidates meet the inclusion and exclusion criteria.

After providing informed consent, eligible patients will undergo a baseline evaluation of PRU levels by means of the VerifyNow system. The research study team will perform the PRU assessment in the cardiovascular research lab as this is considered a research only assessment and is not currently performed as standard of care. Patients with PRU levels ≤208 will undergo cangrelor dose reduction to 0.50 mcg/kg/min, while patients with PRU levels >208 will undergo dose increase to 1.0 mcg/kg/min. At 2 to 12 hours after dose titration, blood samples will be collected for further PD assessment of platelet reactivity. Patients with PRU values >208 will undergo dose increase by 0.25 mc/kg/min up to a maximum of 1.5 mcg/kg/min until a PRU below 208 is achieved, while patients with PRU levels <85 will undergo dose reduction to 0.25 mcg/kg/min, being the lowest possible administration rate allowed during the study period.

Blood sampling for PD testing will be performed at different time points: a) baseline (while on 0.75 mcg/kg/min before dose titration); b) between 2 and 12 hours following dose titration; c) daily (at the same time for the second dose) for up to a maximum of 3 samples after dose titration. 8 ml of blood will be obtained at each time point. Patients receiving an oral P2Y12 inhibitor after the cangrelor infusion start will not undergo further PD testing. All other medications will be prescribed as per standard-of-care prescriptions. Study participation will not interfere with standard clinical treatment or delay care. If cangrelor must be stopped per standard of care prior to study completion, then all collected data will be utilized and study participation will end. At the end of the study participation, the patients will follow the medication regimens prescribed by their treating physician per standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient receiving bridging with standard-dose cangrelor infusion rate of 0.75 mcg/Kg/min for at least two hours as part of their standard of care.
2. Age ≥18 years
3. Provide written informed consent.

Exclusion Criteria:

1. Need for urgent surgery
2. Confirmed or suspected pregnancy (in woman of child-bearing potential) or lactating females
3. Exposure to any oral P2Y12 inhibitor, oral anticoagulant or glycoprotein IIb/IIIa inhibitor within 48 hours.
4. Known allergy, and hypersensitivity, or contraindication to cangrelor, mannitol, sorbitol, or microcrystalline cellulose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-25 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Optimal platelet reactivity | 2-12 hours
  PRU levels between 85 and 208, when using a (PFT)-guided titration of cangrelor infusion rate (cangrelor titration) compared to 0.75 mcg/kg/min (standard-dose infusion) for bridging

SECONDARY OUTCOMES:
Optimal platelet reactivity | 24 hours
  PRU levels between 85 and 208, when using a (PFT)-guided titration of cangrelor infusion rate (cangrelor titration) compared to 0.75 mcg/kg/min (standard-dose infusion) for bridging
Optimal platelet reactivity | 48 hours
  PRU levels between 85 and 208, when using a (PFT)-guided titration of cangrelor infusion rate (cangrelor titration) compared to 0.75 mcg/kg/min (standard-dose infusion) for bridging
Optimal platelet reactivity | 72 hours
  PRU levels between 85 and 208, when using a (PFT)-guided titration of cangrelor infusion rate (cangrelor titration) compared to 0.75 mcg/kg/min (standard-dose infusion) for bridging

CONTACTS AND LOCATIONS:
Overall Officials: Dominick J Angiolillo, MD, PhD, Study Chair — University of Florida College of Medicine - Jacksonville; Luis Ortegra-Paz, MD, PhD, Principal Investigator — University of Florida College of Medicine - Jacksonville

IPD SHARING:
Plan to Share IPD: Yes
Data will be available from the Study Chair upon reasonable request after publication of the main results.
Supporting Information: Study Protocol, Analytic Code